CLINICAL TRIAL: NCT05271149
Title: Effect of Dynamic Orthotic Garment on Foot Pressure Distribution, Postural Control, Functional Performance and Endurance in Spastic Diplegic Cerebral Palsy Children: Randomized Controlled Trial
Brief Title: Dynamic Orthotic Garment in Diplegic Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taibah University (Other)
Responsible Party: Principal Investigator, Hatem Abd Elmohsen Abdel Hamid Emara, Associate professor, Taibah University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Theratog
Record Dates: First submitted 2022-02-21; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Diplegic Cerebral Palsy
Keywords: Theratog; postural control; cerebral palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): conventional physical therapy based on neurodevelopmental techniques, This program will be given for 1 hour, 3 days a week for 12 weeks
  Interventions: Other: Routine Physical Therapy
- study group (Experimental): conventional physical therapy and orthosis (Thera togs) : the child will wear the orthosis for twelve weeks, from 8 to 10 hours a day, during daily-life activities. The child's guardian (mother) will be trained and will receive a DVD recording, with a step-by-step demonstration on the fitting of TheraTogs® in the child. Markings were made in TheraTogs® to facilitate and improve fitting. All necessary support will be offered, with weekly monitoring in person to control the fitting of the orthosis, as well as for possible questions or clarifications.in addition to conventional physical therapy as the control group
  Interventions: Other: Routine Physical Therapy

INTERVENTIONS:
Other: Routine Physical Therapy — Routine physical therapy and orthosis
  Other Names: Experimental: Intervention group

SUMMARY:
This study aims to evaluate the effectiveness of dynamic orthotic garment (Thera togs) on foot pressure distribution, postural control, functional performance and endurance in children with spastic diplegic cerebral palsy (CP). Methods: forty children with spastic diplegic CP, with ages ranging from 8 to 10 years, will be assigned randomly into two groups. The control group will receive the conventional physical therapy, whereas the study group will receive the same program as the control group in addition to Thera togs. Measurement of foot pressure distribution will be performed using a pressure platform, postural control will be evaluated using the trunk control measurement scale Trunk Position Sense pediatric berg balance scale, endurance will be assessed using six-minute walk test (6MWT)

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of dynamic orthotic garment (Thera togs) on foot pressure distribution, postural control, functional performance and endurance in children with spastic diplegic cerebral palsy (CP). Methods: forty children with spastic diplegic CP, with ages ranging from 8 to 10 years, will be assigned randomly into two groups. The control group will receive the conventional physical therapy, whereas the study group will receive the same program as the control group in addition to Thera togs. Measurement of foot pressure distribution will be performed using a pressure platform, postural control will be evaluated using the trunk control measurement scale ,Trunk Position Sense , pediatric berg balance scale, endurance will be assessed using six-minute walk test (6MWT)

ELIGIBILITY:
Inclusion Criteria:

* children with CP who have toe-in gait and had grade 1+ to 2 degree of spasticity according to the Modified Ashworth Scale (MAS) [32]. In addition to score I and II on Gross Motor Function Classification System (GMFCS) scores [33]. As well as the child is required to be able to stand and walk independently.

Exclusion Criteria:

* Children who have impaired hearing or vision, previous lower limb surgery or Botulinum injections of the lower limb muscles within the preceding 6 months will be excluded from the study.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-02-17 (Actual); Primary Completion 2022-05-17 (Estimated); Study Completion 2022-05-20 (Estimated)

PRIMARY OUTCOMES:
Foot pressure distribution | baseline
  Static and dynamic planter pressure measurements to measure peak and mean plantar pressure for each sub-region of the foot (forefoot, mid-foot and rear-foot) expressed in kPa.
Foot pressure distribution | Twelve week
  Static and dynamic planter pressure measurements to measure peak and mean plantar pressure for each sub-region of the foot (forefoot, mid-foot and rear-foot) expressed in kPa.
The trunk control measurement scale | baseline
  to assess the static and dynamic components of trunk control.The minimum score is 1 and the maximum scor is 58.Higher score means better outcome
The trunk control measurement scale | Twelve week
  to assess the static and dynamic components of trunk control .The minimum score is 1 and the maximum scor is 58.Higher score means better outcome
Trunk Position Sense | baseline
  Active position sense of the trunk was assessed using a digital goniometer.
Trunk Position Sense | Twelve weeks
  Active position sense of the trunk was assessed using a digital goniometer.
Pediatric balance scale | baseline
  The Pediatric balance scale, used to determine the dynamic balancing abilities of children with cerebral palsy, shows an excellent inter-rater reliability.The minimum score is 1 and the maximum score is 56.Higher score means better outcome
Pediatric balance scale | Twelve weeks
  The Pediatric balance scale, used to determine the dynamic balancing abilities of children with cerebral palsy, shows an excellent inter-rater reliability.The minimum score is 1 and the maximum score is 56.Higher score means better outcome

SECONDARY OUTCOMES:
Six-minute walk test (6-MWT) | baseline
  distance covered during six minutes will be recorded
Six-minute walk test (6-MWT) | Twelve weeks
  distance covered during six minutes will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Emara, PhD, Principal Investigator — Associate professor
Locations (1):
- Taibah University, Madinah, Almadinah Almunawarah, Saudi Arabia

REFERENCES:
- [Derived] Emara HA, Al-Johany AH, Khaled OA, Al-Shenqiti AM, Ali ARH, Aljohani MM, Sobh E. Effect of the Dynamic Orthotic Garment on Postural Control, and Endurance in Children with Spastic Diplegic Cerebral Palsy: A Randomized Controlled Trial. J Multidiscip Healthc. 2024 Jan 30;17:419-428. doi: 10.2147/JMDH.S438474. eCollection 2024. PMID 38314010